CLINICAL TRIAL: NCT03929328
Title: A Randomized Trial of High Flow Oxygen Therapy in Spontaneous Breathing Trial on Weaning in Mechanical Ventilated Patients.
Brief Title: Effect of High Flow Oxygen Therapy in Spontaneous Breathing Trial on Weaning in Mechanical Ventilated Patients
Acronym: HOST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sang-Min Lee (Other)
Responsible Party: Sponsor-Investigator, Sang-Min Lee, Associate Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOSTLSM2019
Record Dates: First submitted 2019-04-20; First posted 2019-04-26 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Weaning; Mechanical Ventilation; Extubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spontaneous breathing trial with T-piece (No Intervention): Patients were randomized to undergo a spontaneous breathing trial with T-piece that is connected on endotracheal tube. Patients tolerating the spontaneous breathing trial underwent extubation.
- Spontaneous breathing trial with high flow oxygen therapy (Experimental): Patients were randomized to undergo a spontaneous breathing trial with high flow oxygen therapy that is connected on endotracheal tube. Patients tolerating the spontaneous breathing trial underwent extubation.
  Interventions: Procedure: High flow oxygen therapy in spontaneous breathing trial

INTERVENTIONS:
Procedure: High flow oxygen therapy in spontaneous breathing trial — Patients were randomized to undergo a spontaneous breathing trial with high flow oxygen therapy that is connected on endotracheal tube. Patients tolerating the spontaneous breathing trial underwent extubation.
  Arms: Spontaneous breathing trial with high flow oxygen therapy

SUMMARY:
This clinical trial is aimed to show a spontaneous breathing trial using high flow oxygen therapy may lower weaning failure rate and reintubation rate than using T-piece.

DETAILED DESCRIPTION:
We project to test the effect of high flow oxygen therapy in spontaneous breathing trial on weaning in mechanical ventilated patients. Patients will be randomly assigned to undergo a spontaneous breathing trial in one of two ways: with a T-piece therapy or with high flow oxygen therapy. Primary end-points are rate of weaning failure and rate of reintubation within 48 hr of extubation. Weaning failure is defined as failed to spontaneous breathing trial or reintubation within 48 hr of extubation. Secondary end-points are ICU mortality, in-hospital mortality, ICU length of stay, time to reintubation after extubation. Study sample was calculated to detect ability of high flow oxygen therapy to reduce weaning failure from 42 to 15 percent, at two-tailed alpha error of 5% and power of 85% and 98 patients are needed in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or more, both gender
* Receiving endotracheal intubation and mechanical ventilation for more than 12 hours
* Recovery from the precipitating illness
* Weaning readiness according to the following criteria :

  1. Respiratory criteria :

     1. PaO2:FIO2 >150 with FIO2 ≤0.4, PEEP <8 cm H2O
     2. Arterial pH >7.35
     3. Rapid shallow breathing index (RSBI) < 105
     4. Maximum inspiratory pressure (MIP) < -20 cm H20
  2. Clinical criteria :

     1. Absence of electrocardiographic signs of myocardial ischemia
     2. No vasoactive drugs, or vital signs are stable with using vasoactive drugs
     3. Heart rate <140/min,
     4. Hemoglobin >8 g/dL
     5. Temperature <38°C
     6. No need for sedatives, or mental status are stable with sedatives
     7. Presence of respiratory stimulus, and appropriate spontaneous cough
     8. Absence of excessive tracheobronchial secretions

Exclusion Criteria:

* Tracheostomy status
* Decision to stop life-supportive therapies before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of weaning failure | Day 2
  Weaning failure is defined as failed to spontaneous breathing trial or reintubation within 48 hr of extubation

SECONDARY OUTCOMES:
ICU mortality | From the date of randomization until the date of ICU death from any cause, assessed up to 1 month.
  Death in ICU
In-hospital mortality | From the date of randomization until the date of in-hospital death from any cause, assessed up to 3 months.
  Death in hospital
ICU length of stay | Through the study completion, an average of 1 weeks
  Duration in days from day of first spontaneous breathing trial to day of discharge from the ICU
Time to reintubation after extubation | From the date of extubation until the date of reintubation, assessed up to 1 weeks.
  Duration in times from time of extubation to time of reintubation
Rate of reintubation within 48 hr of extubation | Day 2
  Reintubation within 48 hr of extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Min Lee, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Not Provided

REFERENCES:
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Derived] Lee HY, Lee J, Lee SM. Effect of high-flow oxygen versus T-piece ventilation strategies during spontaneous breathing trials on weaning failure among patients receiving mechanical ventilation: a randomized controlled trial. Crit Care. 2022 Dec 23;26(1):402. doi: 10.1186/s13054-022-04281-w. PMID 36564808